CLINICAL TRIAL: NCT06648525
Title: Adebrelimab Combined with Irinotecan Liposomes, 5-fluorouracil, Calcium Folinate ± Lenvatinib As First-line Treatment for Advanced Intrahepatic Cholangiocarcinoma: a Prospective Clinical Study
Brief Title: Adebrelimab Combined with Irinotecan Liposomes, 5-FU, CF ± Lenvatinib As First-line Treatment for Advanced ICC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Zhiwei Li, Head of the gastroenterology ward, Harbin Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-ICC-II-006
Record Dates: First submitted 2024-09-12; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-09

CONDITIONS: Intrahepatic Cholangiocarcinoma (Icc)
Keywords: Adebrelimab; Irinotecan liposomes; Lenvatinib; Intrahepatic Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma; Cirrhosis, Familial, with Pulmonary Hypertension | interventions — lenvatinib; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: Adebrelimab+Irinotecan liposomes+5-fluorouracil+calcium folinate+lenvatinib (Experimental): Adebrelimab in combination with Irinotecan liposomes, 5-fluorouracil, calcium folinate and lenvatinib
  Interventions: Drug: Adebrelimab; Drug: Irinotecan liposomes; Drug: Lenvatinib; Drug: 5-Fluorouracil (5-FU); Drug: Calcium Folinate
- Group B: Adebrelimab+Irinotecan liposomes+5-fluorouracil+calcium folinate (Experimental): Adebrelimab in combination with Irinotecan liposomes, 5-fluorouracil and calcium folinate
  Interventions: Drug: Adebrelimab; Drug: Irinotecan liposomes; Drug: 5-Fluorouracil (5-FU); Drug: Calcium Folinate

INTERVENTIONS:
Drug: Adebrelimab — Adebrelimab, IV
Drug: Irinotecan liposomes — Irinotecan liposomes, IV
Drug: Lenvatinib — Lenvatinib, po
  Arms: Group A: Adebrelimab+Irinotecan liposomes+5-fluorouracil+calcium folinate+lenvatinib
Drug: 5-Fluorouracil (5-FU) — 5-Fluorouracil (5-FU), IV
Drug: Calcium Folinate — Calcium folinate, IV

SUMMARY:
This is a multicenter, open label, randomized, two-arm clinical study to observe and evaluate the efficacy and safety of adebrelimab combined with irinotecan liposomes, 5-fluorouracil, calcium folinate ± lenvatinib as first-line treatment for advanced intrahepatic cholangiocarcinoma (ICC).

DETAILED DESCRIPTION:
This study plans to recruit 68 patients with unresectable ICC who have not received prior systematic treatment. The patients will be randomly divided into two groups. Group A: patients will receive adebrelimab+irinotecan liposomes+5-fluorouracil+calcium folinate+lenvatinib; Group B: patients will receive treatment with adebrelimab+irinotecan liposomes+5-fluorouracil+calcium folinate. The combination of irinotecan liposomes+5-fluorouracil+calcium folinate will be used 9 times (Q2W), and adebrelimab ± lenvatinib will be used until disease progression or medication for 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 75 years old, male or female not limited;
2. Histologically confirmed unresectable locally advanced or metastatic intrahepatic cholangiocarcinoma with measurable tumor lesions (meeting RECIST 1.1 criteria);
3. Have not received systemic anti-tumor treatment in the past;
4. Patients who relapse more than 6 months after curative surgery or after completion of adjuvant therapy (chemotherapy and/or radiotherapy) meet the inclusion criteria;
5. ECOG PS：0-1；
6. Expected survival period ≥ 3 months;
7. The main organ functions are normal, which meets the following criteria:

1) Blood routine examination (without blood transfusion or correction with hematopoietic stimulating factor drugs within 14 days): Hemoglobin (Hb) ≥ 85 g/L; Absolute neutrophil count (ANC) ≥ 1.5 × 109/L; Platelet count (PLT) ≥ 80 × 109/L; 2) Biochemical examination: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 × ULN; Serum total bilirubin (TBIL) ≤ 3 × ULN; Serum creatinine (Cr) ≤ 1.5 × ULN or creatinine clearance rate ≥ 50ml/min; 3) Coagulation function: Activated partial thromboplastin time (APTT), international normalized ratio (INR), prothrombin time (PT) ≤ 1.5 × ULN; 4) Doppler ultrasound evaluation: Left ventricular ejection fraction (LVEF) ≥ 50%; 8. Women of childbearing age must undergo a negative pregnancy test (β HCG) before starting treatment, and women and men of childbearing age (who have sexual relations with women of childbearing age) must agree to continuously use effective contraceptive measures during the treatment period and for 6 months after the last treatment dose; 9. Patients with a history of hepatitis B and C can be included in the study, but active hepatitis B patients must start antiviral therapy before starting the study treatment; 10. Participants voluntarily join the study and sign an informed consent form.

Exclusion Criteria:

1. Pregnant or lactating women, or those who have the ability to conceive but refuse to take contraceptive measures;
2. History of other malignant tumors within the past 5 years, excluding cervical carcinoma in situ or squamous cell carcinoma of the skin that has been adequately treated, or basal cell carcinoma of the skin that has been largely controlled;
3. Merge other serious uncontrolled diseases (such as individuals with a history of difficult to control mental illness or severe intellectual or cognitive impairment; severe heart failure, angina pectoris, myocardial infarction, arrhythmia, etc.);
4. Pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, and severe impairment of lung function;
5. Suffering from active, known or suspected autoimmune diseases. Subjects with hypothyroidism who only require hormone replacement therapy and those with skin diseases that do not require systemic treatment may be included;
6. Easy to bleed, at risk of massive hemoptysis, and with a history of significant coagulation dysfunction;
7. Suffering from hypertension and unable to achieve good control with antihypertensive medication (systolic blood pressure ≥ 140mmHg or diastolic blood pressure ≥ 90mmHg);
8. History of immunodeficiency, including HIV testing positive, having other acquired or congenital immunodeficiency diseases, or having a history of organ transplantation and allogeneic bone marrow transplantation;
9. Severe active infections requiring intravenous antibiotic treatment occur during the screening period;
10. Individuals with multiple factors that affect oral medication (such as inability to swallow, post gastrointestinal resection, chronic diarrhea, and intestinal obstruction);
11. Individuals who are allergic to the experimental drug;
12. Patients who cannot comply with the trial protocol or cooperate with follow-up;
13. The researchers believe that participants should not participate in this experiment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Progression-Free-Survival (PFS) | up to 24 months
  The time from enrollment until tumor progression or death from any cause, whichever occurred first

SECONDARY OUTCOMES:
Objective response rate (ORR) | up to 24 months
  The proportion of patients with a PR or CR, determined by RECIST v1.1 criteria
Disease control rate (DCR) | up to 24 months
  The proportion of patients with a PR, CR, or SD
Overall survival (OS) | up to 24 months
  The time calculated from enrollment until death from any cause, with living patients censored at the last known survival date
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | up to 24 months
  Incidence and severity of adverse events graded according to the NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Harbin Medical University, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No